CLINICAL TRIAL: NCT02212340
Title: Comparison Between Propofol-remifentanil Total Intravenous Anesthesia and Desflurane-remifentanil Balanced Anesthesia With Regard to Post-anesthetic Functional Recovery Measured With QoR-40 in Vitrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3-2014-0104
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Vitrectomy Operation Under General Anesthesia
Keywords: propofol; desflurane; quality of recovery; vitrectomy
MeSH Terms: interventions — Propofol; Remifentanil; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIVA group (Experimental): Anesthesia is maintained with fresofol and remifentanil
  Interventions: Drug: fresofol and remifentanil
- Des group (Active Comparator): Anesthesia is maintained with desflurane and remifentanil
  Interventions: Drug: desflurane and remifentanil

INTERVENTIONS:
Drug: fresofol and remifentanil — Anesthesia is maintained with fresofol and remifentanil in TIVA group or with desflurane and remifentanil in Des group according to randomly allocated group.
  Arms: TIVA group
Drug: desflurane and remifentanil — Anesthesia is maintained with fresofol and remifentanil in TIVA group or with desflurane and remifentanil in Des group according to randomly allocated group.
  Arms: Des group

SUMMARY:
Total intravenous anesthesia (TIVA) and inhalation anesthesia are both widely and safely used, and there are many clinical trials comparing these on various aspects of anesthesia. However, there have not been studies comparing the quality of recovery from the different methods of general anesthesia in vitrectomy. In this study, the investigators compare the functional recovery after general anesthesia in TIVA and inhalation anesthesia with QoR-40 questionnaire in vitrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (20-80 years old) scheduled for vitrectomy surgery undergoing general anesthesia.
2. ASA 1-3

Exclusion Criteria:

1. Patients with allergy to anesthetic agents
2. Anticipated difficult airway
3. BMI > 30 kg/m2
4. Chronic obstructive pulmonary disease
5. Heart failure 6. Unstable angina

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
QoR-40 score | at 6 hours later after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Yonsei University College of Medicine, Seoul, Seoul, South Korea